CLINICAL TRIAL: NCT04486001
Title: COVID-19 Stem Cell Therapy: A Phase I Study of Intravenous Administration of Allogeneic Adipose Stem Cells
Brief Title: Study of Intravenous Administration of Allogeneic Adipose Stem Cells for COVID-19
Acronym: CoronaStem1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Collaborators: VetStem Biopharma, Inc. (Unknown); Fresno Community Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSC-CP-004
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Covid19
Keywords: adipose; stem cell; COVID19; COVID-19; pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Intervention Model Description: single group comparison with cohort of contemporaneous non-treated patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): This is single arm study with only comparison to non-treated cohorts at site.
  Interventions: Biological: PSC-04

INTERVENTIONS:
Biological: PSC-04 — adipose stem cells derived from screened donor lipoaspirate and culture expanded.
  Other Names: allogeneic, adipose-derived stem cells

SUMMARY:
This study is designed rapidly assess safety and preliminary efficacy in hospitalized patients with COVID-19 respiratory distress to provide clinical guidance for possible wider use in treating patients in this pandemic environment. This data will be used for FDA IND filings and pursuit of a BLA.

DETAILED DESCRIPTION:
This study is single arm, non-randomized Phase 1 study of the safety and preliminary efficacy of PSC-04, an adipose-derived allogeneic mesenchymal stem cell. The outcome data will be compared to contemporaneous non-enrolled patients at the same clinical site(s) as the enrolled patients.

Study Objectives:

Primary: To evaluate the safety of intravenous infusion of allogeneic adipose stem cells in patients with COVID-19 disease and respiratory distress.

Secondary: To evaluate a set of secondary safety and efficacy outcome variables to give guidance in assessing the risk/benefit ratio in patients with COVID-19 respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital as in-patient (ward or ICU)
* Respiratory distress - respiratory rate ≥ 30/minute (or PaO2:FiO2 <300)
* Bilateral lung infiltrates (CT or frontal X-ray)
* Supplemental oxygen started but NOT intubated or ventilated
* COVID-19 (SARS-CoV-2) antigen test positive (FDA-approved test);
* CDC confirmation not necessary
* Time from Enrollment to treatment must be less than 24 hours
* Age: 18-80 years
* Gender: any
* Suitability for cellular therapy: In the opinion of the Investigator or the Sponsor the patient is suitable for cellular therapy
* Cognitive function: Able to understand and willing to sign informed consent form or legally authorized representative or surrogate

Exclusion Criteria:

* Intubation / ventilation
* Current therapy is working, and patient is clinically improving
* Disease Conditions: Heart failure severe (NY Heart Association Classification IV); Clinical evidence of left heart failure or volume overload as a primary explanation for the bilateral pulmonary infiltrates; Any disease or condition other than current respiratory COVID-19 disease for which 6-month mortality is estimated to be greater than 50%; Moderate to severe liver failure; Severe chronic respiratory disease or the use of home oxygen use prior to this current illness; Currently receiving extracorporeal life support (ECLS/ECMO)
* Past Disease Conditions: Any history of malignancy within the last 2 years (except for patients in remission or cured of the malignancy); Lung transplant patient or lobectomy; Deep venous thrombosis or pulmonary embolism within past 3 months; History of splenectomy
* Other Experimental Conditions: Currently enrolled or treated in last 60 days in another clinical study
* Consent Issues: Do not resuscitate (DNR) order in place; Not willing to follow lung protective ventilation strategy, if needed
* Concurrent disease or circumstances that Investigator or Sponsor judges to be an unacceptable risk to patient health or a confounding variable to assessment or problem in completion of trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Frequency of all adverse events | Through study completion, an average of three months
  Frequency of all reported adverse events in study
Frequency of infusion related serious adverse events | 6 hours post infusion
  Frequency of SAEs in the 6 hours post-infusion for each infusion
Frequency of serious adverse events | Through study completion, an average of three months
  Frequency of all serious adverse events in study

SECONDARY OUTCOMES:
Mortality | Study days 0-28
  All-cause mortality through Day 28
Ventilator Free Days | Study days 0-28
  Ventilator free days through Study day 28
ICU Free Days | Days 0 through 28
  Total days not in ICU from Study day 0 through Study day 28
Total Hospital Days | Days 0 through discharge, an average of 28 days
  Total Days in Hospital from Day 0 through discharge for survivors
Total ICU Days | Days 0 through discharge, an average of 28 days
  Total Days in ICU from Day 0 through discharge for survivors
Improvement in Oxygenation | Study days 0, 2, 4, 6
  Improvement in oxygenation comparing Study day 0, to days 2, 4, 6

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD JD, Study Director — Sorrento Therapeutics, Inc.
Locations (1):
- Fresno Community Hospital, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rogers CJ, Harman RJ, Bunnell BA, Schreiber MA, Xiang C, Wang FS, Santidrian AF, Minev BR. Rationale for the clinical use of adipose-derived mesenchymal stem cells for COVID-19 patients. J Transl Med. 2020 May 18;18(1):203. doi: 10.1186/s12967-020-02380-2. PMID 32423449